CLINICAL TRIAL: NCT00464711
Title: Brain GABA Levels and Treatment Response in Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, David Mischoulon, M.D., Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001295
Record Dates: First submitted 2007-04-23; First posted 2007-04-24 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
Keywords: depression; biology
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escitalopram (Other): single arm
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Dose determined per clinical discretion. All participants begin on 10mg po qd of escitalopram, and can increase the dose to 30mg po qd over the 12 weeks of the study.
  Other Names: Lexapro

SUMMARY:
This study will evaluate changes in brain gamma-aminobutyric acid (GABA) levels due to treatment with escitalopram in people with major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a severe form of depression. MDD can significantly interfere with an individual's thoughts, behavior, mood, and physical health. People who suffer from MDD often experience feelings of worthlessness; they may feel hopeless and may be unable to cope with problems in their life. In addition, they often experience sleep disruption, loss of appetite, and chronic pain.

The purpose of the study is to compare images taken of the brains of people who are depressed and the brains of healthy volunteers. Specifically, we want to see if symptoms of depression are related to a decrease in a brain chemical called GABA. We measure the concentration of GABA using a brain-scanning device called "magnetic resonance spectroscopy" (or "MRS"), which is a type of MRI.

The study lasts for 14 weeks and involves 8 visits to our MGH clinic in Boston. The first visit is the screening visit, which can last up to 3 hours. The rest of the visits are about a half hour long and take place every other week. In addition to these 8 visits, there are also 2 visits to McLean Hospital Brain Imaging Center for the MRS scans. The first scan takes place within a few days after the screening visit, and the second scan will be at the end of the 14 weeks. Each scan visit lasts between an hour and a half and two hours. Subjects are reimbursed $50 per MRS scan and $25 per visit to McLean to cover travel costs.

All subjects in this study will receive escitalopram (or Lexapro), which is an antidepressant medication approved by the Food and Drug Administration. Subjects start at 10 mg daily of the escitalopram, but may be increased up to 30 mg if the study doctor thinks it is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic criteria for current Major Depressive Disorder
* Men or women aged 18-65
* Medication-free for one week prior to the start of the study
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Anyone who is suicidal
* Pregnant or breastfeeding women
* Anyone with a serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* Anyone with a history of seizure disorder or hypothyroidism
* Anyone with a history of psychiatric disorders including bipolar disorder, schizophrenia, psychoses, or substance abuse (including alcohol abuse active within the last 12 months)
* Anyone with a history of intolerance or multiple adverse drug reactions or allergy to (es)citalopram.
* Patients who are currently taking medications active on GABA, including benzodiazepines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Iosifescu, MD, Principal Investigator — Depression Clinical and Research Program, Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Massachusetts General Hospital Depression Clinical and Research Program Website — http://www.massgeneral.org/depression/

RESULTS

PARTICIPANT FLOW:
Groups:
- Escitalopram: 40 subjects met inclusion/exclusion criteria and started treatment with escitalopram
Period: Overall Study
Arm/Group | Escitalopram
Started | 40
Completed | 25
Not Completed | 15

BASELINE CHARACTERISTICS:
Groups:
- Escitalopram: 40 subjects met inclusion/exclusion criteria and started study treatment
Arm/Group | Escitalopram
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.675 (14.08)
Gender [Count of Participants; unit: Participants]
  Female | 21
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Response and Remitter Status at Endpoint, Based on Change in Depression Severity Rating Scores
Description: The primary outcome in this study was based on the Hamilton Rating Scale for Depression, 17 items (HAMD-17). Clinical Response status was defined as > 50 % reduction in HAMD-17 scores from baseline to endpoint. Clinical Remitter status was defined as endpoint HAMD-17 score < 8.
  40 patients (21 female) with major depressive disorder (MDD) started the 12 week study treatment with escitalopram, 25 patients (15 female) completed the 12 weeks.
Time Frame: 12 weeks
Population: 40 patients (21 female) with MDD enrolled in the 12 week study, 25 patients (15 Female) completed. Current analyses are based on completers only.
Measure: Number; unit: participants
Groups:
- Open Label Escitalopram: All subjects were treated with open label escitalopram
Arm/Group | Open Label Escitalopram
Number analyzed (Participants) | 25
participants
  Clinical Response | 16
  Clinical Remission | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 12 weeks of treatment.
Arm/Group | Escitalopram
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 20/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=40)
Insomnia (General disorders) | 9 (9)
GI Upset (Gastrointestinal disorders) | 8 (8) — GI upset category includes GI upset, nausea, diarrhea, Gas, stomach cramps, indigestion
Fatigue/Sedation (General disorders) | 5 (5)
Headache (General disorders) | 4 (4)
Sexual Side Effects (General disorders) | 4 (4) — Sexual side effects included reports of general sexual side effects, decreased sex drive, anorgasmia, and erectile dysfunction.
Jitteriness/Agitation (General disorders) | 2 (2)
Decreased Appetite (General disorders) | 2 (2)
Increased sweatiness (General disorders) | 2 (2)
Increased Appetite (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No